CLINICAL TRIAL: NCT05870085
Title: Impact of Neuro-linguistic Programs on the Academic Performance of Primary School Students in Lebanon: Triggers, Attention Deficit Hyperactivity Disorder Symptoms and Their Effect on Behavior and Academic Performance of Schoolchildren
Brief Title: Impact of Neuro-linguistic Programming on Schoolchildren's Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Georges Hatem, Clinical Professor, Lebanese University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 3/23/D
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Academic Skill Disorder; Child Behavior
MeSH Terms: conditions — Learning Disabilities; Child Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Neuro-linguistic program — Intervention: Neuro-linguistic program developed by three specialists (a clinical psychologist, a social worker, and one education specialist).
  4 (45 minutes) sessions for teachers, and 2 for children (total of 6 sessions)

SUMMARY:
Neuro-Linguistic Programming (NLP) is a methodology developed in the 1970s by Richard Bandler and John Grinder, based on the idea that language and behavior are interconnected and can be systematically modeled and changed. NLP is often used as a form of psychotherapy, coaching, or personal development, although its effectiveness has been debated in the scientific community.

NLP practitioners believe that our thoughts, emotions, and behavior are influenced by our internal representations of the world, which are constructed through language and sensory experiences. Changing the use of language and the perception of experiences, thoughts, emotions, and behavior can be adjusted accordingly. NLP uses various techniques to achieve this, including reframing, anchoring, and rapport-building. Reframing involves changing the perception of a situation by putting it in a different context or perspective. Anchoring consists in associating a particular state of mind or emotion with a specific physical or sensory stimulus, such as a touch or a smell. Rapport-building involves establishing a connection and a sense of trust with another person through mirroring and matching their body language, tone of voice, and language patterns.

DETAILED DESCRIPTION:
Neuro-Linguistic Programming (NLP) techniques have been used in various contexts, including education. Some educators and practitioners believe that NLP can help children develop their communication skills, self-confidence, and self-awareness and improve their learning outcomes. Some NLP techniques adapted for children include: (1) Anchoring involves linking a particular emotional or sensory state with a physical stimulus, such as a touch or a visual cue. For example, a teacher might use a specific gesture or word to help a child feel more confident before a test. (2) Reframing: This technique involves helping a child see a situation or problem differently. For example, a teacher might help a child reframe a difficult math problem as a fun challenge. And (3) Meta-modeling: This technique involves helping children become more aware of their language patterns and the language patterns of others, which can improve communication skills and self-awareness.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren aged between 5 and 11 years attending the same school for at least a year.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Identification of school triggers through ''Identify School Triggers'' questionnaire | 2 months after the intervention
  130 children will be asked to fill out the ''Identify school triggers'' questionnaire by rating items depending on the strength of the trigger impact. A score over 20 will be calculated and the strength of the triggers will be evaluated after categorizing the scores.
Schoolchildren's strengths and difficulties progression through the Strengths and Difficulties Questionnaire | 2 months after the intervention
  A parent (mother or father or legal guardian) of 130 children will be asked to fill out a survey. The first 25 items in the SDQ comprise 5 scales of 5 items each. It is usually easiest to score all 5 scales before working out the Total Difficulties score. Somewhat True is always scored as 1, but the scoring of Not True and Certainly True varies with each item. For each of the 5 scales, the score can range from 0-10 if all 5 items were completed. Scale scores can be prorated if at least 3 items were completed. Using the comments, a "substantial risk of clinically significant problems" score on the Total Difficulties Score can be used to identify likely ''cases" with mental disorders.
Concentration, hyperactivity, and reasoning of schoolchildren through the Vanderbilt Assessment Scale | 2 months after the intervention
  Two different teachers will complete the survey for each student (130 students and 12 teachers). The initial assessment scales, parent and teacher, have two components:
  Symptom assessment and impairment in performance. Symptom assessment screens for symptoms that meet the criteria for inattentive (items 1-9) and hyperactive attention deficit hyperactivity disorder (ADHD) (items 10-18). To meet the requirements for the diagnosis, one must have at least six positive responses to either the inattentive nine or hyperactive nine core symptoms, or both. The specific item sets and numbers of positives required for each co-morbid symptom screen set are detailed below. The second section of the scale has many performance measures, scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.

CONTACTS AND LOCATIONS:
Overall Officials: Roula Abou Assi, PhD, Study Director — Lebanese University
Locations (1):
- Notre dame de la paix, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No